CLINICAL TRIAL: NCT03569033
Title: A Phase 2a, Randomized, Placebo-Controlled Clinical Trial to Evaluate the Efficacy, Safety and Tolerability of MK-7264 on Acute Cough in Participants With Induced Viral Upper Respiratory Tract Infection
Brief Title: Study of Gefapixant (MK-7264) in Acute Cough for Participants With Induced Viral Upper Respiratory Tract Infection (URTI) (MK-7264-013)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The data did not support study endpoints for acute cough, based on an interim efficacy analysis; not due to safety concerns.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7264-013; MK-7264-013 (Other: Merck Protocol Number); 2017-000472-28 (EudraCT Number)
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Results first posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-11

CONDITIONS: Acute Cough
MeSH Terms: interventions — Gefapixant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Gefapixant 45 mg BID (Experimental): Participants will receive a gefapixant 45 mg tablet twice daily (BID) for 7 days.
  Interventions: Drug: Gefapixant
- Placebo BID (Placebo Comparator): Participants will receive a matching placebo tablet BID for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gefapixant — Gefapixant 45 mg will be administered orally.
  Other Names: MK-7264
  Arms: Gefapixant 45 mg BID
Drug: Placebo — Placebo tablet matching gefapixant will be administered orally.
  Arms: Placebo BID

SUMMARY:
The purpose of the study is to evaluate the efficacy, safety, and tolerability of gefapixant (MK-7264) in adult participants with induced viral upper respiratory tract infections (URTI).

ELIGIBILITY:
Inclusion Criteria:

* In good general health
* Susceptible to human rhinovirus type 16 (HRV-16)
* Male or non-pregnant and non-breast feeding female
* If female of reproductive potential, agrees to use 1 form of acceptable birth control

Exclusion Criteria:

* Donated blood within 56 days or donated plasma within 7 days prior to dosing
* History of significant multiple and/or severe allergies
* Recent history of respiratory tract infection
* History of cancer
* Body mass index <18 kg/m^2 or ≥40 kg/m^2
* History of major surgery or loss of 1 unit of blood
* History of allergic reaction to sulfonamides
* Received medications within 14 days prior to randomization
* Significantly abnormal laboratory tests at Screening
* Current smoker, smoked within 5 years of Screening, or significant past smoking history
* History of alcohol or drug abuse

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2018-07-04 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Hvivo Service Limited. Queen Mary BioEnterprises ( Site 0003), London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Smith JA, Kitt MM, Bell A, Noulin N, Tzontcheva A, Seng MM, Lu S. Treatment with the P2X3-Receptor Antagonist Gefapixant for Acute Cough in Induced Viral Upper Respiratory Tract Infection: A Phase 2a, Randomized, Placebo-Controlled Trial. Pulm Ther. 2022 Sep;8(3):297-310. doi: 10.1007/s41030-022-00193-w. Epub 2022 Aug 15. PMID 35969360

RESULTS

PARTICIPANT FLOW:
Groups:
- Gefapixant 45 mg BID: Participants received a gefapixant 45 mg tablet twice daily (BID) for 7 days.
- Placebo BID: Participants received a matching placebo tablet BID for 7 days.
Period: Overall Study
Arm/Group | Gefapixant 45 mg BID | Placebo BID
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gefapixant 45 mg BID | Placebo BID | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.9 (7.4) | 24.3 (5.6) | 24.6 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 19 | 19 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 21 | 21 | 42
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Awake Coughs Per Hour on Day 3
Description: Awake cough frequency (coughs per hour) was assessed by an objective digital cough-counting device (VitaloJAK™ cough monitor) on Day 3.
Time Frame: Day 3
Population: All randomized participants who received at least 1 dose of trial intervention and had confirmation of viral shedding at 72 hours post inoculation with human rhinovirus type 16 (HRV-16)
Measure: Least Squares Mean (95% Confidence Interval); unit: Coughs per hour
Arm/Group | Gefapixant 45 mg BID | Placebo BID
Number analyzed (Participants) | 23 | 19
Coughs per hour | 2.38 [1.01 to 3.75] | 2.70 [1.21 to 4.19]
Statistical Analysis 1: Comparison: Gefapixant 45 mg BID vs Placebo BID; Test type: Other; p = 0.748, Longitudinal Data Analysis; Difference in Least Squares Means = -0.32, 95% CI 2-sided [-2.29 to 1.66]

2. Secondary Outcome: Change From Baseline in the Cough Severity Visual Analog Scale (VAS) Score on Day 3
Description: The Cough Severity VAS was scored from 0 to 100 using a 100 mm visual analogue scale. Participants were asked to mark on a 100 mm scale between 0 (no cough) and 100 (the worst cough severity). Cough VAS was evaluated at Baseline and on Day 3.
Time Frame: Baseline and Day 3
Population: All randomized participants who received at least 1 dose of trial intervention and had confirmation of viral shedding at 72 hours post inoculation with HRV-16
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Gefapixant 45 mg BID | Placebo BID
Number analyzed (Participants) | 23 | 19
Scores on a scale | 6.07 [1.79 to 10.35] | 5.08 [0.39 to 9.78]
Statistical Analysis 1: Comparison: Gefapixant 45 mg BID vs Placebo BID; Test type: Other; p = 0.754, ANCOVA; Difference in Least Squares Means = 0.99, 95% CI 2-sided [-5.33 to 7.30]

3. Secondary Outcome: Change From Baseline in the Mean Total Daily Cough Severity Diary (CSD) Score on Day 3
Description: The Mean Total Daily CSD Score is calculated using the daily CSD instrument, a 7-item, disease-specific, patient-reported outcome measure with a recall period of "today" (the current day). The measure evaluates frequency of cough (3 items); intensity of cough (2 items); and disruption due to cough (2 items). Each of these 7 items is rated on an 11-point scale, ranging from 0 (best) to 10 (worst), with higher scores indicating greater severity. The total daily CSD score is the sum of these 7 item scores (Min=0, Max=70). The Mean Total Daily CSD Score (the sum of these 7 item scores divided by 7) was calculated at Baseline and on Day 3.
Time Frame: Baseline and Day 3
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Gefapixant 45 mg BID | Placebo BID
Number analyzed (Participants) | 23 | 19
Scores on a scale | 2.71 [0.46 to 4.97] | 1.91 [-0.55 to 4.38]
Statistical Analysis 1: Comparison: Gefapixant 45 mg BID vs Placebo BID; Test type: Other; p = 0.627, ANCOVA; Difference in Least Squares Means = 0.80, 95% CI 2-sided [-2.50 to 4.10]

4. Secondary Outcome: Change From Baseline in the Leicester Cough Questionnaire (LCQ)-Acute Score on Day 3
Description: The LCQ-Acute is a 19-item health-related quality-of-life (HRQoL) questionnaire specific for acute cough which contains three domains (i.e., physical, psychological, and social). It is calculated as a mean score for each domain ranging from 1 to 7, and total score ranging from 3 to 21. Each item on the LCQ-acute assesses symptoms or the impact of symptoms on HRQoL in the last 24 hours using a 7-point Likert scale ranging from 1 to 7. Higher scores indicate better HRQoL. Participants' perception of their cough severity was assessed, based on the LCQ-Acute score, at Baseline and on Day 3.
Time Frame: Baseline and Day 3
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Gefapixant 45 mg BID | Placebo BID
Number analyzed (Participants) | 23 | 19
Scores on a scale | -0.26 [-0.51 to -0.01] | -0.35 [-0.62 to -0.08]
Statistical Analysis 1: Comparison: Gefapixant 45 mg BID vs Placebo BID; Test type: Other; p = 0.631, ANCOVA; Difference in Least Squares Means = 0.09, 95% CI 2-sided [-0.28 to 0.45]

5. Secondary Outcome: Percentage of Participants Who Experienced One or More Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a study participant administered a pharmaceutical product that does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Time Frame: Up to 21 days
Population: All randomized participants who received at least 1 dose of study treatment
Measure: Number; unit: Percentage of participants
Arm/Group | Gefapixant 45 mg BID | Placebo BID
Number analyzed (Participants) | 23 | 23
Percentage of participants | 100 | 95.7

6. Secondary Outcome: Percentage of Participants Who Discontinued Treatment Due to an Adverse Event (AE)
Description: as for outcome 5
Time Frame: Up to Day 7
Population: All randomized participants who received at least 1 dose of study treatment
Measure: Number; unit: Percentage of participants
Arm/Group | Gefapixant 45 mg BID | Placebo BID
Number analyzed (Participants) | 23 | 23
Percentage of participants | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Up to 21 days
Description: All randomized participants who received at least 1 dose of study treatment
Groups:
- MK-7264 45 mg BID: Participants received a gefapixant 45 mg tablet BID for 7 days.
- Placebo: Participants received a matching placebo tablet BID for 7 days.
Arm/Group | MK-7264 45 mg BID | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 23/23 | 22/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-7264 45 mg BID (N=23) | Placebo (N=23)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 2 (2) | 0 (0)
Medical device site erythema (General disorders) | 16 (16) | 17 (17)
Upper respiratory tract infection (Infections and infestations) | 20 (20) | 21 (22)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (10) | 0 (0)
Hypogeusia (Nervous system disorders) | 3 (5) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated because the data did not support study endpoints for acute cough, based on an interim efficacy analysis; not due to safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the sponsor, the investigator agrees to submit all manuscripts or abstracts to the sponsor before submission. This allows the sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT03569033/Prot_SAP_000.pdf